CLINICAL TRIAL: NCT07318701
Title: Multi-agent Large Language Models for Multidisciplinary Decision Support in Cervical Cancer During Pregnancy
Brief Title: Multi-agent LLMs for Decision Support in Cervical Cancer During Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Keqin Hua, Doctor, Principal Investigator, Clinical Professor, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-33
Record Dates: First submitted 2025-12-18; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer
Keywords: Large Language Model; Cervical cancer during pregnancy; Multi-agent
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: multi-disciplinary agents group (Experimental): generate diagnosis and treatment opinions from multi-disciplinary agents
  Interventions: Other: multi-disciplinary agents group
- Arm2: real MDT group/ junior doctors group/junior doctors after referring to agent results group (Placebo Comparator): generate diagnosis and treatment opinions from real MDT group/ junior doctors group/junior doctors after referring to agent results group
  Interventions: Other: real MDT group; Other: junor doctor group; Other: junor doctor group with aid of MDT agents

INTERVENTIONS:
Other: multi-disciplinary agents group — generate diagnosis and treatment opinions for each case from multi-disciplinary agents
  Arms: Arm1: multi-disciplinary agents group
Other: real MDT group — generate diagnosis and treatment opinions for each case from a real MDT team inclduing senior physicians from relevant departments, including gynecologic oncology, pediatrics, obstetrics, medical oncology and radiation oncology.
  Arms: Arm2: real MDT group/ junior doctors group/junior doctors after referring to agent results group
Other: junor doctor group — generate diagnosis and treatment opinions for each case from junior doctor who are residents from relevant departments, including gynecologic oncology, pediatrics, obstetrics, medical oncology and radiation oncology.
  Arms: Arm2: real MDT group/ junior doctors group/junior doctors after referring to agent results group
Other: junor doctor group with aid of MDT agents — generate diagnosis and treatment opinions for each case from junior doctor who are residents from relevant departments, including gynecologic oncology, pediatrics, obstetrics, medical oncology and radiation oncology after referring to the results from MDT agent .
  Arms: Arm2: real MDT group/ junior doctors group/junior doctors after referring to agent results group

SUMMARY:
The aim of this study is to develop an AI-assisted decision-making system based on multi-agent large language models and to evaluate its effectiveness and accuracy in the diagnosis and treatment of cervical cancer during pregnancy.

DETAILED DESCRIPTION:
This project intends to construct China's first artificial intelligence model for the vertical field of "multidisciplinary team (MDT) consultation" for cervical cancer during pregnancy. Centered on the massive case data of gynecological oncology from Obstetrics and Gynecology Hospital of Fudan University, combined with cervical cancer during pregnancy guidelines to formulate multi-oncology department judgment standards, it will focus on overcoming key technical bottlenecks such as model reliability, model result evaluation, and multi-agent collaborative scheduling. With this model as the engine, a trinity AI hub will be built, driven by agent collaboration and combined with a guideline-based evaluation system to realize intelligent support for " cervical cancer during pregnancy MDT consultation + guideline evaluation". By constructing a vertical model for MDT consultation for cervical cancer during pregnancy, MDT AI agent consultation, and a guideline-based evaluation system, the project will comprehensively improve the standardization, homogenization level and efficiency of diagnosis and treatment, promote the upgrading of the diagnosis and treatment capabilities for cervical cancer during pregnancy diagnosis and treatment capabilities, and provide more accurate and high-quality medical service guarantees for patients.

1. Vertical Large Language Model Based on the guidelines for cervical cancer during pregnancy and other relevant authoritative guidelines and expert consensus, it provides high-quality structured knowledge support and reliable decision-making explanation basis for the gynecological oncology vertical model.

   Construct a high-quality gynecological oncology vertical corpus: Address the difficulty of manual corpus construction, build controllable data generation based on the existing full tumor process, establish a gynecological oncology corpus with high accuracy and strong generalization ability, and enhance the quality of fine-tuning data.

   Construct a vertical gynecological oncology large language model: Improve the basic professional capabilities of the model through methods such as maximizing internal coherence and measuring mutual predictability; introduce a length penalty mechanism and neighborhood-adaptive reinforcement learning based on large language models to enable the language model to discriminate gynecological oncology logic. Through a reference reward mechanism based on standard answers, the gynecological guideline reward model supports the reinforcement learning of the gynecological model and solves the key problem of model interpretability. Improve core clinical tasks such as early screening, accurate staging diagnosis, personalized treatment plan recommendation, risk stratification assessment and intelligent follow-up of gynecological tumors, achieve or exceed the level of international advanced similar models in key performance indicators, and provide scientific and reliable intelligent support for clinical diagnosis and treatment decisions.
2. Agent Construction Construct a collaborative intelligent platform driven by exclusive diagnosis and treatment agents for each department: With hierarchical modular design as the core and agent cluster as the driving force, it covers the full-cycle diagnosis and treatment process of cervical cancer during pregnancy. The underlying data layer integrates clinical business data and specialized knowledge bases to support the diverse AI capabilities of the model layer; the Agent framework layer, as the technical hub, realizes multi-model scheduling, long-term and short-term memory management, and automatic arrangement of diagnosis and treatment processes through modules such as model gateway, memory enhancement, and strategy orchestration; the platform management layer provides visual scenario configuration, rule engine and workflow management to ensure medical compliance; the application layer includes gynecological oncology, neonatology, chemotherapy, and obstetrics agents to form a collaborative network. Design task routing and time-sharing classification scheduling strategies, assign tasks based on Agent capabilities and load, prioritize quality control and auxiliary diagnosis and treatment tasks, and improve computing power efficiency; realize the full life cycle management of Agents, including registration, release, and optimization, configure vertical model binding, prompts, etc., optimize corpus quality through user feedback, and coordinate the division of labor among multiple Agents through workflow engine to solve problems such as dynamic branches of complex diagnosis and treatment paths and knowledge tool collaboration, ensuring efficient collaboration.

   Construct the platform's intelligent scheduling and management capabilities for Agents: Design task routing to assign tasks based on Agent capabilities and current load; statistically analyze Agent usage efficiency and frequency to design execution priorities, and improve the efficiency of computing resource utilization. Design time-sharing classification scheduling strategies based on the confidence interval of AI in clinical business and the feasibility priority of non-core process substitution. Provide independent deployment capabilities for core businesses to avoid computing resource contention, ensure scheduling executability, and improve business resilience.
3. Guideline-Based MDT Decision Evaluation System Analyze and restructure knowledge based on the Guidelines for cervical cancer during pregnancy, extract key diagnosis and treatment points applicable to MDT, and establish an exclusive evaluation index system covering gynecological oncology, obstetrics, chemotherapy, and neonatology to quantitatively evaluate and compare diagnosis and treatment plans from different sources.

In real case datasets, we will retrospectively enrolled patients diagnosed as cervical cancer during in obstetrics and gynecology hospital from January 2007 to December 2025. The inclusion criteria is as follows: 1) Pathologically confirmed diagnosis of cervical cancer; 2) Confirmed intrauterine pregnancy status via ultrasound. 3) Patients receiving initial treatment. 4)Agreement to participate in the study with signed informed consent. The exclusion criteria is as follows: 1) Previous treatment received for cervical cancer during pregnancy. 2) Pathological pregnancy states (e.g., ectopic pregnancy). 3) Inability or unwillingness to provide signed informed consent. For each case, we will collect diagnosis and treatment opinions from multi-disciplinary agents, junior doctors, and junior doctors after referring to agent results respectively. Then we calculate and compare accuracy and consistency scores according to evaluation indicators of each discipline for the three parties' results.

In virtual case datasets, similar to criteria for the retrospective study section, 100 virtual cases of cervical cancer during pregnancy were generated. These cases were randomly divided in a 1:1 ratio into MDT-agents group and a real MDT team group. We will calculate accuracy and compare results according to the same evaluation indicators. Besides, we will also compare the consuming time for each case by MDT-agents and real MDT team respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of cervical cancer.
2. Confirmed intrauterine pregnancy status via ultrasound.
3. Patients receiving initial treatment.
4. Agreement to participate in the study with signed informed consent.

Exclusion Criteria:

1. Previous treatment received for cervical cancer during pregnancy.
2. Pathological pregnancy states (e.g., ectopic pregnancy).
3. Inability or unwillingness to provide signed informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the MDT decision | immediately after the intervention
  scores, from 0 to 100, accuracy of the MDT decision according to evaluation indicators of each discipline

SECONDARY OUTCOMES:
Consuming time | immediately after the intervention
  seconds, consuming time for generating MDT decisions from MDT agents/ real MDT team

CONTACTS AND LOCATIONS:
Overall Officials: Keqin Hua, Doctor, Principal Investigator — Gynecology and obstetrics hospital of fudan university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li R, Wang X, Berlowitz D, Mez J, Lin H, Yu H. CARE-AD: a multi-agent large language model framework for Alzheimer's disease prediction using longitudinal clinical notes. NPJ Digit Med. 2025 Aug 24;8(1):541. doi: 10.1038/s41746-025-01940-4. PMID 40849361
- [Result] Meyer R, Hamilton KM, Truong MD, Wright KN, Siedhoff MT, Brezinov Y, Levin G. ChatGPT compared with Google Search and healthcare institution as sources of postoperative patient instructions after gynecological surgery. BJOG. 2024 Jul;131(8):1154-1156. doi: 10.1111/1471-0528.17746. Epub 2024 Jan 4. No abstract available. PMID 38177090
- [Result] Patel JM, Hermann CE, Growdon WB, Aviki E, Stasenko M. ChatGPT accurately performs genetic counseling for gynecologic cancers. Gynecol Oncol. 2024 Apr;183:115-119. doi: 10.1016/j.ygyno.2024.04.006. Epub 2024 Apr 26. PMID 38676973
- [Result] Hermann CE, Patel JM, Boyd L, Growdon WB, Aviki E, Stasenko M. Let's chat about cervical cancer: Assessing the accuracy of ChatGPT responses to cervical cancer questions. Gynecol Oncol. 2023 Dec;179:164-168. doi: 10.1016/j.ygyno.2023.11.008. Epub 2023 Nov 21. PMID 37988948
- [Result] Garg P, Mohanty A, Ramisetty S, Kulkarni P, Horne D, Pisick E, Salgia R, Singhal SS. Artificial intelligence and allied subsets in early detection and preclusion of gynecological cancers. Biochim Biophys Acta Rev Cancer. 2023 Nov;1878(6):189026. doi: 10.1016/j.bbcan.2023.189026. Epub 2023 Nov 20. PMID 37980945
- [Result] Bedi S, Jain SS, Shah NH. Evaluating the clinical benefits of LLMs. Nat Med. 2024 Sep;30(9):2409-2410. doi: 10.1038/s41591-024-03181-6. No abstract available. PMID 39060659
- [Result] Macchia G, Ferrandina G, Patarnello S, Autorino R, Masciocchi C, Pisapia V, Calvani C, Iacomini C, Cesario A, Boldrini L, Gui B, Rufini V, Gambacorta MA, Scambia G, Valentini V. Multidisciplinary Tumor Board Smart Virtual Assistant in Locally Advanced Cervical Cancer: A Proof of Concept. Front Oncol. 2022 Jan 3;11:797454. doi: 10.3389/fonc.2021.797454. eCollection 2021. PMID 35047408
- [Result] Amant F, Berveiller P, Boere IA, Cardonick E, Fruscio R, Fumagalli M, Halaska MJ, Hasenburg A, Johansson ALV, Lambertini M, Lok CAR, Maggen C, Morice P, Peccatori F, Poortmans P, Van Calsteren K, Vandenbroucke T, van Gerwen M, van den Heuvel-Eibrink M, Zagouri F, Zapardiel I. Gynecologic cancers in pregnancy: guidelines based on a third international consensus meeting. Ann Oncol. 2019 Oct 1;30(10):1601-1612. doi: 10.1093/annonc/mdz228. PMID 31435648
- [Result] Peccatori FA, Azim HA Jr, Orecchia R, Hoekstra HJ, Pavlidis N, Kesic V, Pentheroudakis G; ESMO Guidelines Working Group. Cancer, pregnancy and fertility: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi160-70. doi: 10.1093/annonc/mdt199. Epub 2013 Jun 27. No abstract available. PMID 23813932
- [Result] Halaska MJ, Drochytek V, Shmakov RG, Amant F. Fertility sparing treatment in cervical cancer management in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2021 Sep;75:101-112. doi: 10.1016/j.bpobgyn.2021.03.014. Epub 2021 Apr 22. PMID 33992541